CLINICAL TRIAL: NCT06512948
Title: Early Surgical Effects and Influencing Factors of High Tibial Osteotomy in the Treatment of Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Shufeng Li (Other)
Responsible Party: Sponsor-Investigator, Shufeng Li, Chief Physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: 0000-0001-6044-0655
Record Dates: First submitted 2024-01-04; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Logistics regression model: This article is a retrospective study, which mainly incorporates patients' preoperative and postoperative imaging parameters and demographic data into Logistics regression analysis to analyze factors that may affect the surgical effect. No interventions such as medication are involved.
  Interventions: Procedure: High tibial osteotomy

INTERVENTIONS:
Procedure: High tibial osteotomy — Surgical treatment for patients with osteoarthritis and indications for high tibial osteotomy

SUMMARY:
Exploring the factors influencing postoperative functional recovery after high tibial osteotomy

DETAILED DESCRIPTION:
A retrospective study was conducted on patients who underwent HTO at the First Affiliated Hospital of Shandong First Medical University from January 2018 to December 2020, and the preoperative and postoperative imaging indicators [medial proximal tibial angle (MPTA), joint line intersection angle (JLCA), hip-knee-ankle angle (HKA angle), knee weight-bearing line percentage (WBL%), postoperative distraction distance, postoperative distraction angle] and knee joint function score [including the American Hospital for Special Surgery (HSS) knee score, American Knee Society score (KSS), Lysholm score, Western Ontario and McMaster Universities Osteoarthritis Index score (WOMAC), and all were included in logistic regression analysis to study the surgical effect and impact of HTO factor

ELIGIBILITY:
Inclusion Criteria:

* Medial knee OA, varus deformity is mainly in the tibia
* Aged ≤70 years old, with higher requirements for future activities
* Knee joint extension is limited to ≤10°, and flexion is >90°
* Body Mass Index (BMI) ≤ 40
* No subchondral bone wear

Exclusion Criteria:

* There is a history of fracture or surgery of the lower limb on the operated side
* Traumatic KOA
* Combined with nerve, muscle or connective tissue diseases
* Incomplete imaging data and loss of follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study subjects were patients who underwent medial open HTO for KOA at the First Affiliated Hospital of Shandong First Medical University from January 2018 to December 2020. This article included a total of 45 patients with grade II and grade III according to the Kellgren-Lawrence arthritis classification. There were 28 cases, including 5 grade IV patients.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Imaging parameters | an average of 1 year after the surgery
  Medial proximal tibial angle
Imaging parameters | an average of 1 year after the surgery
  Opening gap
Imaging parameters | an average of 1 year after the surgery
  the weight bearing line ratio
Imaging parameters | an average of 1 year after the surgery
  joint line convergence angle
Imaging parameters | an average of 1 year after the surgery
  Hip-knee-ankle
Imaging parameters | an average of 1 year after the surgery
  opening angle

SECONDARY OUTCOMES:
function score | an average of 1 year after the surgery
  the US Hospital for special surgery knee-rating score
function score | an average of 1 year after the surgery
  American knee society knee score
function score | an average of 1 year after the surgery
  Lysholm
function score | an average of 1 year after the surgery
  Western Ontario and McMaster Universities Osteoarthritis Index

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Zhao, professor, Study Director — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No